CLINICAL TRIAL: NCT05920382
Title: Radiofrequency Ablation for the Treatment of Post-knee Arthroplasty Chronic Pain. A Randomized Double-blind Study. A Novel Approach.
Brief Title: Radiofrequency Ablation for the Treatment of Post-knee Arthroplasty Chronic Pain.
Acronym: CSAPG-37
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Principal Investigator, Italo Pisani, Head of Pain Unit, Consorci Sanitari de l'Alt Penedès i Garraf
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSAPG-37
Record Dates: First submitted 2023-05-30; First posted 2023-06-27 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Chronic Post-surgical Pain; Chronic Post Operative Pain; Chronic Knee Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized double-blind clinical trial with two arms:
  Radiofrequency Arm (RFA): Thermal radiofrequency will be applied to the sensory nerves of the knee, along with local anesthetic and corticosteroid infiltration.
  Control Arm (CA): Simulated radiofrequency will be applied to the sensory nerves of the knee, along with local anesthetic and corticosteroid infiltration.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The assessment of the results will be carried out by personnel hired for this purpose, who will be unaware of the patient's group allocation. Similarly, neither the investigators nor the collaborators present on the day of the intervention will be aware of the results of the applied technique. The data analysts will also be blinded to the study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency arm (Experimental): After identifying the nerves to be treated via ultrasound and confirming with neurostimulation, 1 ml of 2% lidocaine will be administered, followed by radiofrequency ablation. The physical parameters used are as follows: 90 seconds, 80 degrees Celsius, with a 22g needle with an active tip of 10 mm.
  Interventions: Procedure: Radiofrequency ablation of peripheral nerves.
- Control arm (Sham Comparator): In the same manner as with the RF group, the nerves to be treated are identified via ultrasound and confirmed by neurostimulation. Subsequently, sham radiofrequency is performed for 90 seconds.
  Interventions: Procedure: Radiofrequency ablation of peripheral nerves.

INTERVENTIONS:
Procedure: Radiofrequency ablation of peripheral nerves. — Randomized double-blind clinical trial where we will apply thermal radiofrequency to the sensory terminal branches of the femoral nerve in the knee, including the vasto medial nerve, vasto lateral nerve, vasto intermedio nerves, and the infrapatellar branch of the saphenous nerve.
  Other Names: Radiofrecuency arm; Sham arm

SUMMARY:
Knee osteoarthritis pain is one of the conditions commonly seen in general and specialized medicine. Knee arthroplasty is one of the most successful orthopedic surgeries for the treatment of this disease, significantly improving pain, disability, and the overall quality of life for patients who undergo it. However, there is a subgroup of individuals in whom the pain persists or even worsens. Radiofrequency has been introduced over 10 years ago as a neuroablative technique targeting the genicular nerves, which innervate the sensory terminals of the knee joint, for the treatment of chronic pain in that region before or after arthroplasty. However, the results have not been entirely consistent. Recent anatomical studies have demonstrated the presence of other sensory terminal branches of the femoral nerve, such as the infrapatellar branch of the saphenous nerve, medial vastus nerve, intermediate vastus nerve, and lateral vastus nerve, which could be useful targets for the treatment of post-knee arthroplasty pain. To date, no studies have been conducted to address post-knee arthroplasty pain through the application of thermal radiofrequency on the sensory branches of the knee from the femoral nerve (infrapatellar branch of the saphenous nerve, medial vastus nerve, intermediate vastus nerve, lateral vastus nerve). Therefore, The investigators aim to conduct a randomized double-blind clinical trial where The investigators will apply thermal radiofrequency on the sensory terminal branches of the femoral nerve in the knee, based on recent anatomical studies. The objective of the study is to determine if radiofrequency ablation of sensory nerves in the knee improves pain and disability in patients with post-knee arthroplasty chronic pain at the L'Alt Penedés-Garraf Health Consortium. Method: This is a randomized double-blind clinical trial with two arms. Two groups will be used, where one group will receive thermal radiofrequency of sensory nerves in the knee, and the other group will receive a placebo treatment. The hypothesis The investigators propose is that radiofrequency ablation will alleviate at least 50% of baseline pain and disability in at least 50% of the patients.

DETAILED DESCRIPTION:
Degenerative knee osteoarthritis pain is one of the main reasons for consultation in general and specialized medicine. Its assessment and treatment impose a high cost on healthcare systems, accounting for 0.5% of Spain's gross domestic product. Given the magnitude of the disease and the disability it causes in affected individuals, multiple therapies have been proposed, ranging from pharmacological therapy with nonsteroidal anti-inflammatory drugs, opioids, antidepressants, capsaicin cream treatment, and physiotherapy, to intra-articular treatments with corticosteroids and viscosupplements like hyaluronic acid, platelet-rich plasma, etc. Knee arthroplasty is one of the most successful orthopedic surgeries in current medicine, significantly improving pain, disability, and the overall quality of life for patients who undergo it. However, postoperative pain following knee arthroplasty remains a challenging problem, with incidence rates of pain and disability after the procedure ranging from 48% to 34%, respectively, at 3 and 6 months post-surgery, with iatrogenic nerve injury being the most common cause. There are limited therapeutic alternatives available from this point onwards.

Since the first description of using radiofrequency for the treatment of intractable chronic pain, it has become not only a tool for pain management but also a cornerstone in pain units' treatment. The use of radiofrequency ablation for pain is based on the premise that the transmission of radiofrequency current near nociceptive pathways would interrupt the pain stimulus through the destruction of the nervous tissue. Thermal radiofrequency has been successfully used in the treatment of facetogenic low back pain, sacroiliac joint pain, and discogenic low back pain.

In the year 2011, the first study was conducted on radiofrequency of the sensory nerves of the knee, known as the genicular nerves, using femoral and tibial condyles as anatomical references and fluoroscopy as an imaging guide. Unfortunately, discrepancies in terminology and anatomical descriptions have led to confusion among interventional physicians. Other researchers have demonstrated discrepancies with the studies published in 2011, making it more difficult to standardize the technique of neuroablation of these nerves. More recently, other researchers demonstrated a specific anatomical-ultrasound correlation of sensory terminal branches of the femoral and sciatic nerves that innervate the knee. The involved nerves include the infrapatellar branch of the saphenous nerve, the nerve to the medial vastus muscle, the nerve to the intermediate vastus muscle, the nerve to the lateral vastus muscle, the anterior branch of the obturator nerve, the recurrent peroneal nerve, and the lateral retinacular nerve.

Study justification:

Post-knee arthroplasty pain remains an unresolved problem, with various techniques applied to different anatomical targets yielding inconsistent results. To date, no studies have addressed post-knee arthroplasty pain through the application of thermal radiofrequency on sensory branches of the femoral nerve, namely the infrapatellar branch of the saphenous nerve, nerve to the medial vastus muscle, nerve to the intermediate vastus muscle, and nerve to the lateral vastus muscle guided by ultrasound.

Therefore, The investigators propose to conduct a randomized double-blind clinical trial where The investigators will apply thermal radiofrequency on the sensory terminal branches of the knee from the femoral nerve, including the medial vastus nerve, lateral vastus nerve, intermediate vastus nerve, and infrapatellar branch of the saphenous nerve.

Hypothesis:

Patients who receive radiofrequency ablation would experience a percentage reduction of at least 50% in baseline pain and disability at 3 months, which The investigators consider a clinically significant effect.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have undergone knee arthroplasty.
* Chronic knee pain post-knee arthroplasty for at least 6 months after the procedure and less than 5 years.
* Pain intensity on the numerical visual scale ≥ 5 out of 10 points.
* Stable pain for the last 30 days.
* The knee is the location with the highest intensity of pain, in the case of patients with multiple joint pains.

Exclusion Criteria:

* Acute knee pain.
* Psychiatric illness or dementia that may interfere with or hinder study assessments.
* Diagnosis of fibromyalgia, chronic fatigue syndrome, or central sensitization syndrome.
* Knee infiltration with corticosteroids in the past 30 days.
* Changes in oral analgesic medication in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change Pain and Disability measured by Western Ontario and McMaster Universities Arthritis Index, (WOMAC). | 3 month
  Determine if radiofrequency ablation of the medial vastus nerve, infrapatellar branch of the saphenous nerve, intermediate vastus nerve, and lateral vastus nerve improves pain and disability at 3 months compared to baseline, as measured by WOMAC questionnaire, in patients with post-knee arthroplasty pain, compared to patients treated with placebo.
  The WOMAC test consists of several questions that address different aspects related to pain and functionality of the affected joint. These questions are divided into three main domains:
  Pain, Stiffness, Physical function The change in test scores will be evaluated throughout the study period, comparing them to the baseline.

SECONDARY OUTCOMES:
Changes in pain measured by the Numeric Rating Scale for pain. (NRS) | 3 month
  Determine whether radiofrequency ablation of the sensory nerves in the knee under study improves pain at 3 months compared to baseline in patients with post-knee arthroplasty pain, compared to patients treated with placebo.
  It consists of a straight line or a series of numbers from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable." The change in test scores will be evaluated throughout the study period, comparing them to the baseline.
Neuropathic pain measured by Neuropathic Pain questionnaire (DN4) | 3 month
  Determine if radiofrequency ablation of the studied knee sensory nerves improves pain at 3 months compared to baseline in patients with neuropathic pain following knee arthroplasty, compared to patients treated with placebo.
Depression and anxiety measured by Hospital Anxiety and Depression Scale (HADS) | 3 month
  Measure levels of depression and anxiety in patients undergoing radiofrequency ablation and study their influence on the response to radiofrequency therapy of the studied knee sensory nerves. The scores on the HADS are interpreted as follows:
  Anxiety:
  0-7: Normal (no clinically significant anxiety) 8-10: Mild anxiety 11-14: Moderate anxiety 15-21: Severe anxiety
  Depression:
  0-7: Normal (no clinically significant depression) 8-10: Mild depression 11-14: Moderate depression 15-21: Severe depression
Degree of satisfaction with the procedure performed measured by categorical satisfaction scale of our hospital's pain unit. | 3 month
  Compare the level of satisfaction among patients undergoing radiofrequency ablation of the knee sensory nerves for the treatment of chronic post-knee arthroplasty pain.
  Not satisfied: The treatment provided no relief and worsened my pain. Slightly satisfied: The treatment had minimal results and my pain barely improved.
  Moderately satisfied: The treatment had moderate results and my pain improved to some extent.
  Quite satisfied: The treatment was effective and my pain improved significantly.
  Very satisfied: The treatment was highly effective and my pain completely disappeared.
Safety from the applied treatment measured by number of adverse events associated with the technique. | 3 month
  Determine the safety of radiofrequency ablation of the knee sensory nerves in terms of the number of adverse events associated with the technique.
Duration (YEARS) of pain and treatment outcomes measured by Numeric Rating Scale for pain. | 3 month
  Assess if the time measured in years since the last knee arthroplasty is related to the outcomes of the applied therapy, such as the 50% reduction in pain and disability measured by the visual numeric pain scale.
Duration (YEARS) of pain and treatment outcomes measured by WOMAC questionnaire. | 3 month
  Assess if the time measured in years since the last knee arthroplasty is related to the outcomes of the applied therapy, such as the 50% reduction in pain and disability measured by WOMAC questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: JOSEP M SEGUR, PHD, Study Director — BARCELONA UNIVERSITY
Locations (1):
- Consorci Sanitari Alt'Pènedes i Garraf, Barcelona, Catalonia, Spain